CLINICAL TRIAL: NCT05473390
Title: Effect of FES of Back Muscles on Spinal Posture and Gait in Hemiplegia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mohammed Youssef Elhamrawy, Principal Investigator, Beni-Suef University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: on posture & Balance
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): 20 patient with hemiplegia
  Interventions: Other: functional electrical stimulation; Other: kinesotaping
- control group (Active Comparator): 20 patient with hemiplegia
  Interventions: Other: functional electrical stimulation

INTERVENTIONS:
Other: functional electrical stimulation — functional electrical stimulation on back muscles
Other: kinesotaping — no intervention
  Arms: study group

SUMMARY:
Hemiplegic patient have unbalanced posture because paralysis leads to muscle atrophy, which then causes an unbalanced alignment in the structure of spinal joints. Evaluation and therapy of postural alignment are important as early predictable factors in the overall daily function of stroke patients

DETAILED DESCRIPTION:
To evaluate whether the application of FES of the back muscles in hemiplegic affect spinal posture and/or gait

ELIGIBILITY:
Inclusion Criteria:

* 20 children with c.p. hemiplegia
* moving and performing daily activities independently
* no problems in terms of verbal communication
* no physical and cognitive restrictions.

Exclusion Criteria:

* Having cognitive impairment as tested by the Mini-Mental State Examination (with scores < 24)
* Uncontrolled hypertension (systolic blood pressure > 160 mmHg)
* Joint replacement
* Incontinence

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
spinal posture | "up to 8 weeks"
  3 D assessment of spinal posture using Microsoft kinect
Balance assessment | "up to 8 weeks"
  balance assessment using Time up and go test TUG high risk (>13.5 seconds): ____ None/low/moderate: (<13.5 seconds) and Berg scale normal score for elderly (45:56)

CONTACTS AND LOCATIONS:
Overall Officials: mohammed s Saif, phd, Principal Investigator — National institute for Gerontology
Locations (1):
- National institute for Gerontology, Cairo, Egypt